CLINICAL TRIAL: NCT04084574
Title: Diet and Hypertension Management in African Americans With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00102823
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Diseases; High Blood Pressure
Keywords: Racial disparities; Hypertension; Diet; Kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Diet Counseling (Experimental): Groups of 4-6 participants will attend 12 weekly dietitian-led counseling sessions and receive coaching on practical strategies to enhance DASH diet adherence and reduce daily sodium intake.
  Interventions: Behavioral: DASH diet counseling
- Standard of Care (Other): Participants will meet one-on-one with the study dietitian for a single 30- minute encounter and be advised to limit daily sodium intake per current clinical practice guidelines for hypertension in patients with CKD. Educational handouts and tip sheets about practical strategies to reduce dietary sodium will be distributed.
  Interventions: Behavioral: DASH diet counseling

INTERVENTIONS:
Behavioral: DASH diet counseling — Culturally-appropriate, disease-sensitive counseling intervention to enhance DASH diet adherence in Blacks with CKD compared to standard of care condition

SUMMARY:
The purpose of this study is to determine cultural and disease-related barriers and facilitators to following the Dietary Approaches to Stop Hypertension (DASH) dietary pattern among Black Americans with moderate chronic kidney disease (CKD) and test the impact of a behavioral diet counseling intervention on DASH diet adherence, blood pressure, and CKD-relevant outcomes.

DETAILED DESCRIPTION:
Excess cardiovascular disease (CVD) mortality among Black Americans with CKD is a significant US public health disparity. Compared to their White counterparts, Blacks develop CKD earlier in life and Blacks with CKD are 3 times more likely to progress to kidney failure necessitating dialysis or kidney transplantation, and are 1.5 times more likely to die prematurely from CVD. Hypertension, which is also more prevalent, more severe, and less often controlled in Blacks with CKD compared to Whites, is a leading cause of CKD and CVD, and a major contributor to the racial disparity in CVD mortality. Thus, improving hypertension in Blacks with CKD could have a profound positive impact on an important minority health issue.

The DASH diet lowers BP and reduces CVD risk in patients with hypertension and has a greater effect on BP in Blacks compared to Whites. However, the effect of the DASH diet on BP in Blacks with CKD has not been established. First, investigators will conduct a qualitative study to identify self-perceived barriers and facilitators of DASH diet adherence among Blacks with moderate CKD. Then, investigators will conduct feasibility, acceptability, and preliminary efficacy testing of a disease-sensitive, culturally-appropriate diet counseling intervention on DASH adherence and blood pressure in Blacks with CKD.

Prior to the clinical trial portion of this project Qualitative Focus Groups were held to identify self-perceived barriers and facilitators of DASH diet adherence among African Americans with CKD. Three to 4 groups of 6-8 participants were asked semi-structured questions to determine self-perceived sociocultural barriers and facilitators of DASH diet adherence and disease-specific factors that may influence their ability and willingness to follow a DASH-style diet. The information in the rest of this record pertains to the clinical trial portion of the project.

ELIGIBILITY:
Inclusion Criteria:

* Black race (self-identified)
* ≥21 years old
* CKD defined as an eGFR of 30-59 ml/min/1.73m2

Exclusion Criteria:

* History of kidney transplant
* Pregnant of breast-feeding
* Risk factors for hyperkalemia including insulin-dependent diabetes mellitus, diabetes with poor blood glucose control (A1C >10), baseline serum potassium ≥4.8 mg/dl, and serum bicarbonate <18 mg/dl
* History of hypertension in the preceding 6 months defined as serum potassium greater than 5.1 mg/dl
* Risk for hypotension or severe hypertension (SBP <120 or ≥180 or DBP ≥110 mmHg)
* History of kidney transplant
* Lack of English language proficiency

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Tyson, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be available to other researchers

REFERENCES:
- [Background] Tyson CC, Davenport CA, Lin PH, Scialla JJ, Hall R, Diamantidis CJ, Lunyera J, Bhavsar N, Rebholz CM, Pendergast J, Boulware LE, Svetkey LP. DASH Diet and Blood Pressure Among Black Americans With and Without CKD: The Jackson Heart Study. Am J Hypertens. 2019 Sep 24;32(10):975-982. doi: 10.1093/ajh/hpz090. PMID 31187128
- [Background] Tyson CC, Barnhart H, Sapp S, Poon V, Lin PH, Svetkey LP. Ambulatory blood pressure in the dash diet trial: Effects of race and albuminuria. J Clin Hypertens (Greenwich). 2018 Feb;20(2):308-314. doi: 10.1111/jch.13170. Epub 2018 Jan 31. PMID 29384243
- [Background] Tyson CC, Lin PH, Corsino L, Batch BC, Allen J, Sapp S, Barnhart H, Nwankwo C, Burroughs J, Svetkey LP. Short-term effects of the DASH diet in adults with moderate chronic kidney disease: a pilot feeding study. Clin Kidney J. 2016 Aug;9(4):592-8. doi: 10.1093/ckj/sfw046. Epub 2016 Jun 5. PMID 27478603
- [Background] Tyson CC, Kuchibhatla M, Patel UD, Pun PH, Chang A, Nwankwo C, Joseph MA, Svetkey LP. Impact of Kidney Function on Effects of the Dietary Approaches to Stop Hypertension (Dash) Diet. J Hypertens (Los Angel). 2014;3:1000168. doi: 10.4172/2167-1095.1000168. PMID 26380159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients at a single academic medical center were recruited by invitation via their electronic patient portal or mailed letter.
Pre-assignment Details: Of 204 individuals who completed the pre-screening survey, 158 were eligible for further screening, 86 consented to the study, and 31 met final inclusion criteria and were randomized to the intervention or control group.
Period: Overall Study
Arm/Group | Behavioral Diet Counseling | Standard of Care
Started | 16 | 15
Completed | 13 | 15
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Relocated out of state | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Diet Counseling | Standard of Care | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (6.7) | 72.7 (6.2) | 71.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 15 | 31
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Group Counseling Sessions Attended by Participants Randomized to the Treatment Arm
Time Frame: Up to 12 weeks
Population: Only relevant to the Behavioral Diet Counseling arm.
Measure: Mean (Standard Deviation); unit: sessions per participant
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 16 | 0
sessions per participant | 8.9 (4.2) |

2. Primary Outcome: Number of Participants Who Completed Data Collection Visits at Scheduled Study Timepoints
Description: Number of randomized participants who provided blood and urine biospecimens, clinic and 24-hour ambulatory blood pressure measurements, and 24-hour dietary recall data during scheduled data collection visits at baseline, 1 month, 3 months, and 6 months.
Time Frame: Baseline, 1 month, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 16 | 15
Participants
  Baseline | 16 | 15
  1 month | 14 | 15
  3 months | 14 | 14
  6 months | 13 | 15

3. Primary Outcome: Change in 24-hour Mean Systolic Blood Pressure
Description: Change was measured by determining the difference in 24-hr mean systolic blood pressure (mmHg) obtained at 12 weeks (end of treatment) from baseline value.
Time Frame: Baseline to 12 weeks
Population: Data not collected on 3 participants in the Behavioral Diet Counseling arm and 4 participants in the Standard of Care arm.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 13 | 10
mmHg | -0.9 (16.1) | 4.0 (9.1)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 0.3968, t-test, 2 sided — The threshold for statistical significance is p = 0.05; Mean Difference (Net) = -4.9, 95% CI 2-sided [-16.8 to 6.9], Standard Deviation 13.5 — Between group difference in mean blood pressure change from baseline for Standard of Care group minus Behavioral Diet Counseling group

4. Primary Outcome: Change in Serum Potassium Concentration
Description: Change was measured by determining the difference in serum potassium at 12 weeks (end of treatment) from baseline value.
Time Frame: Baseline to 12 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 14 | 14
mmol/L | 0.06 (0.46) | 0.01 (0.53)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 0.07926, t-test, 2 sided; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.33 to 0.44], Standard Deviation 0.50 — Between group difference from baseline for Standard of Care group minus Behavioral Diet Counseling group

5. Primary Outcome: Change in 24 Hour Urine Sodium Concentration
Description: Change was measured by determining the difference in 24 hour urine sodium concentration at 12 weeks (end of treatment) from baseline value.
Time Frame: Baseline to 12 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: mmol/L/day
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 14 | 14
mmol/L/day | -8.2 (37.1) | -19.9 (75.3)

6. Primary Outcome: Change in 24 Hour Urine Sodium Concentration
Description: as for outcome 5
Time Frame: Baseline to 12 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: mmol/L/day
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 14 | 14
mmol/L/day | -8.2 (37.1) | -19.9 (75.25)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 0.0673, t-test, 2 sided; Mean Difference (Net) = 11.7, 95% CI 2-sided [-34.2 to 58.6], Standard Deviation 59.3

7. Primary Outcome: Change in 24 Hour Urine Phosphorus Concentration
Description: Change was measured by determining the difference in 24 hour urine phosphorus concentration at 12 weeks (end of treatment) from baseline value.
Time Frame: Baseline to 12 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: mg/dL/day
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 14 | 14
mg/dL/day | -73.0 (180.9) | -62.3 (197.3)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 0.8821, t-test, 2 sided; Mean Difference (Net) = -10.7, 95% CI 2-sided [-157.8 to 136.4], Standard Deviation 189.3 — Between group difference from baseline for Standard of Care group minus Behavioral Diet Counseling group

8. Primary Outcome: Change in 24 Hour Urine Urea Nitrogen Concentration
Description: Change was measured by determining the difference in 24 hour urine urea nitrogen concentration at 12 weeks (end of treatment) from baseline value.
Time Frame: Baseline to 12 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 14 | 14
mcg/mL | -0.5 (2.5) | -1.07 (3.9)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 0.6479, t-test, 2 sided; Mean Difference (Net) = 0.6, 95% CI 2-sided [-2.0 to 3.1], Standard Deviation 3.3 — Between group difference from baseline for Standard of Care group minus Behavioral Diet Counseling group

9. Secondary Outcome: Change in Clinic Mean Systolic Blood Pressure
Description: Change was measured by determining the difference in clinic mean systolic blood pressure (mmHg) obtained at 12 weeks (end of treatment) from baseline value.
Time Frame: Baseline to 12 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 14 | 14
mmHg | 4.6 (21.5) | -2.4 (22.2)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 0.4044, t-test, 2 sided; Mean Difference (Net) = 7.0, 95% CI 2-sided [-10.0 to 24.0], Standard Deviation 21.8 — Between group difference in mean blood pressure change from baseline for Behavioral Diet Counseling group minus Standard of Care group

10. Secondary Outcome: Change in Body Weight
Description: Change was measured by determining the difference in body weight obtained at 12 weeks (end of treatment) from baseline value.
Time Frame: Baseline to 12 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 14 | 14
kg | 0.16 (1.65) | -1.18 (3.76)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 0.2374, t-test, 2 sided; Mean Difference (Net) = 1.34, 95% CI 2-sided [-0.97 to 3.60], Standard Deviation 2.91

11. Secondary Outcome: Change in Mean Clinic Systolic Blood Pressure From 12 Weeks (End of Treatment) to 24 Week Observation
Description: Change was measured by determining the difference in mean clinic systolic blood pressure (mmHg) obtained at 24 weeks from 12 weeks.
Time Frame: 12 weeks to 24 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 13 | 13
mmHg | -7.9 (13.9) | -5.2 (13.3)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 0.6188, t-test, 2 sided; Mean Difference (Net) = -2.69, 95% CI 2-sided [-13.71 to 8.33], Standard Deviation 13.62 — Between group difference from 12 weeks to 24 weeks for Behavioral Diet Counseling group minus Standard of Care group

12. Secondary Outcome: Change in Body Weight From 12 Weeks (End of Treatment) to 24 Week Observation
Description: Change was measured by determining the difference in body weight obtained at 24 weeks from 12 weeks.
Time Frame: 12 weeks to 24 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 13 | 13
kg | -0.77 (1.97) | 0.62 (1.62)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 0.0546, t-test, 2 sided; Mean Difference (Net) = -1.39, 95% CI 2-sided [-2.82 to 0.03], Standard Deviation 1.79 — Between group difference from 12 weeks to 24 weeks for Behavioral Diet Counseling group minus Standard of Care group

13. Secondary Outcome: Change in DASH Diet Score From 12 Weeks (End of Treatment) to 24 Week Observation
Description: Change was measured by determining the difference in DASH diet score obtained at 24 weeks from 12 weeks. The DASH score, ranging from 8 to 40 points with eight components, focuses on food and nutrients for managing hypertension. The eight components are "fruits", "vegetables", "nuts and legumes", "whole grains", "low-fat dairy", "sodium", "red and processed meats", and "sweetened beverages". A higher score indicates better diet quality.
Time Frame: 12 weeks to 24 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 12 | 12
score on a scale | 0.25 (1.41) | 0.25 (1.00)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 1.00, t-test, 2 sided; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.98 to 0.98], Standard Deviation 1.20 — Between group difference from 12 weeks to 24 weeks for Behavioral Diet Counseling group minus Standard of Care group

14. Secondary Outcome: Change in DASH Diet Score From Baseline to 12 Weeks (End of Treatment)
Description: as for outcome 13
Time Frame: Baseline to 12 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Diet Counseling | Standard of Care
Number analyzed (Participants) | 13 | 13
score on a scale | 0.15 (1.26) | -0.14 (1.69)
Statistical Analysis 1: Comparison: Behavioral Diet Counseling vs Standard of Care; Test type: Superiority; p = 1.00, t-test, 2 sided; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.89 to 1.49], Standard Deviation 1.50

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Behavioral Diet Counseling | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 4/16 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Behavioral Diet Counseling (N=16) | Standard of Care (N=15)
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 — Serum creatinine >30% at previous visit or occurrence of adverse event involving 'acute kidney injury'
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 1 — Serum potassium 5.1-5.5 mmol/L
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 — Serum potassium 5.6-5.9 mmol/L

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT04084574/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT04084574/ICF_000.pdf